CLINICAL TRIAL: NCT03418402
Title: Post Operative Pain After Laparoscopic Hysterectomy Using Airseal® Versus Standard Insufflation System: A Randomized Prospective Study
Brief Title: Post Operative Pain After Laparoscopic Hysterectomy Using Airseal® Versus Standard Insufflation System
Acronym: AIRSEAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-27; 2017-A01640-53 (Registry Identifier: ID RCB)
Record Dates: First submitted 2018-01-18; First posted 2018-02-01 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Laparoscopic Hysterectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Airseal® (Experimental): Low pression laparoscopy with a 8 to 10 mmHg pneumoperitoneum.
  Interventions: Device: Airseal®
- Standard insufflator (Active Comparator): laparoscopy realised with our usual insufflation system and a 12 to 15 mmHg pneumoperitoneum.
  Interventions: Device: Standard insufflator

INTERVENTIONS:
Device: Airseal® — Total laparoscopic hysterectomy: Approach according to the Open-Laparoscopy technique and use of the insufflation system.
  Arms: Airseal®
Device: Standard insufflator — Standard insufflator
  Arms: Standard insufflator

SUMMARY:
Airseal® is an insufflation management system for laparoscopic surgery which provides stable pneumoperitoneum, continuous smoke evacuation and valve-free access to the abdominal cavity. It allows an optimal exposure with a low-pression pneumoperitoneum, which is rarely possible with our standard insufflation system under a pneumoperitoneum of 12 millimetres of mercury(mmHg).

The objective of this study is to compare the use of Airseal® system with a low pression pneumoperitoneum and our standard insufflation system usually used in our center in term of postoperative abdominal pain after laparoscopic hysterectomy for benign disease.

This superiority prospective randomized trial is designed to include all patients > 18 years old referred for laparoscopic total hysterectomy for benign disease (with or without uni or bilateral annexectomy). Each patient would be randomized to one of this two following groups :

* " Airseal® " group : use of AIRSEAL® to obtain stable low pression laparoscopy with a 8 to 10 mmHg pneumoperitoneum.
* " Standard laparoscopy " group : laparoscopy realised with our usual insufflation system and a 12 to 15 mmHg pneumoperitoneum.

The primary end point is mean intensity of abdominal pain six hours after the end of surgery (H6), measured by simple numerical scale (ENS).

The secondary end points are:

* peroperative endpoints : operative time, blood loss, use of additional ways of increasing exposure, peroperative complications, conversion to laparotomy, feeling of the surgeon regarding the difficulty of the surgery (measured by a simple numerical scale)
* early postoperative endpoints : intensity of abdominal pain at the entry in recovery room (H0), at twelve hours after the end of surgery (H12), twenty four hours (H24) and forty eight hours (H48) ; intensity of scapular pain at the same times (H0, H6, H12, H24 and H48), need for analgesic administration (regarding to the standardized analgesic protocol), difference in the hemoglobin level before surgery and the first day after, early postoperative complications, necessity of a second surgery and the reason, length of hospital stay.
* late postoperative end points : estimated time to return to optimal quality of life, global satisfaction of patients evaluated by the Quality Of Life Questionnaire Short Form 12.

It will be estimate that the use of Airseal® will reduce the mean abdominal pain at H6 post operative of 1 point on the simple numerical scale compared to our standard insufflation system, with a standard deviation of 1,5. Type 1 and 2 errors were set to the usual levels of 0,05 and 0,20 respectively (power of 80%). Assuming a 10% withdrawal rate, the sample size would be 80 patients (40 patients in each group).

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 18 years old.
* Patients who agreed to participate in the study and signed informed consent.
* Surgical indication by laparoscopy of total interadnexal hysterectomy or associated with unilateral or bilateral adnexectomy, for benign pathology, without any other associated surgical procedure.
* Absence of contraindications to the taking of analgesics provided for in the standardized protocols of analgesia per and post-operative.

Exclusion Criteria:

* Patients at least 18 years old.
* Patients who agreed to participate in the study and signed informed consent.
* Surgical indication by laparoscopy of total interadnexal hysterectomy or associated with unilateral or bilateral adnexectomy, for benign pathology, without any other associated surgical procedure.
* Absence of contraindications to the taking of analgesics provided for in the standardized protocols of analgesia per and post-operative.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-02-08 (Actual); Primary Completion 2020-06-11 (Actual); Study Completion 2020-07-08 (Actual)

PRIMARY OUTCOMES:
Assessment of pain by simple numerical scale | six hours
  The primary end point is mean intensity of abdominal pain measured by simple numerical scale. a score of 0 to 10 best describes the importance of the patient's pain. The score 0 corresponds to "no pain". Note 10 is the maximum "pain" imaginable

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Olivier ARNAUD, Director, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France